CLINICAL TRIAL: NCT03834337
Title: Characteristics of Patients With Symptomatic Active Neurocysticercosis and Effect of Treatment on Symptoms, Lesions and Quality of Life in Resource-poor Rural Areas of Eastern Africa - TOPANA, a Multi-centre Prospective Cohort Study.
Brief Title: Treatment of Patients With Active Neurocysticercosis in Eastern Africa
Acronym: TOPANA
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); University of Zambia (Other); Sokoine University of Agriculture (Other)
Responsible Party: Sponsor
Other Study IDs: TOPANA
Record Dates: First submitted 2019-01-30; First posted 2019-02-07 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Neurocysticercosis
MeSH Terms: conditions — Neurocysticercosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multi-centre prospective cohort study of symptomatic patients with active neurocysticercosis (NCC) aims to identify factors related to treatment success of anthelmintic therapy.

Neurological symptom/sign and cyst resolution, quality of life, accuracy and performance of serological T. solium diagnostics and NCC-specific immunological parameter will be followed up at multiple time points in the study. The final assessment will be done six months after the end of anthelmintic treatment. This study aims to guide treatment of NCC in sub-Saharan Africa by identifying factors that are associated with treatment outcomes.

The factors that cause some people to fail complete resolution of all cysts and/or symptoms/signs are unknown.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be included who
* Meet the definitions of active NCC
* Have epilepsy, epileptic seizures or chronic/severe progressive headaches
* Are physically and mentally fit enough for treatment
* Are willing to be hospitalized and to receive the standard treatment for NCC
* Are willing to participate a follow-up for six months
* Are willing and able to consent to this study, with consent recorded on a signed consent form

Exclusion Criteria:

* Potential participants who will not meet the above inclusion criteria will be excluded.
* Women who are pregnant will not be included, but re-evaluated for inclusion into the study after they have given birth.
* Potential participants who are currently taking or have taken albendazole, praziquantel, or a corticosteroid within the past 12 months will be excluded.
* People with uncontrolled hypertension and/or diabetes will be excluded from the study but will be re-evaluated for inclusion once their hypertension and/or diabetes have been treated.
* People with chronic consuming illness such as cancer and those with mental handicap severe enough to not allow them to follow the study instructions or reliably take their medication will be excluded.
* Children aged <10 years.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with active, symptomatic neurocysticercosis in rural areas in Tanzania and Zambia
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Resolution of lesions | Change in number of active cysts from before treatment to six months after treatment termination
  The number of active cysts identified by CT scan after treatment
Symptom/sign frequency | Change of symptom/sign frequency from before treatment to six months after treatment termination
  The percentage of participants who exhibit a neurological symptom/sign of NCC: chronic/severe progressive headache or epileptic seizures.

SECONDARY OUTCOMES:
Health-related Quality of Life (all patients): WHOQOL-Bref questionnaire | Change in quality of life from before treatment to six months after treatment termination
  The change in participants' self-reported quality of life from before to after treatment, as measured by the WHOQOL-Bref questionnaire (in all participants) [World Health Organization Quality of Life questionnaire; consisting of 26 items].
  Quality of life is assessed by four domains - physical health, psychological, social relationships and environment. In each domain a score of 0 to 100 can be achieved. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). Domains are not summarised to an overall score.
Health-related Quality of Life (epileptic patients) | Change in quality of life from before treatment to six months after treatment termination
  The change in participants' self-reported quality of life from before to after treatment, as measured by the QOLIE-31 questionnaire [Quality of life in epilepsy - 31 items].
  The score consists of 7 domains which all are range from 0 to 100%. Those domains are: seizure worry, overall quality of life, emotional well-being, energy/fatigue, cognitive, medication effects, social function. The seven domains are then summarized to an overall score by applying weights to each category. The overall score ranges from 0 to 100% with 100% being best possible quality of life.
Change in presence of T.solium-specific antigen | Change in presence of T.solium-specific antigen from before treatment to six months after treatment termination
  Change in presence of T.solium-specific antigen in the blood of patients with active neurocysticercosis

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Medical Research, Dar es Salaam, Tanzania

REFERENCES:
- [Result] Stelzle D, Makasi C, Schmidt V, Trevisan C, Van Damme I, Ruether C, Dorny P, Magnussen P, Zulu G, Mwape KE, Bottieau E, Prazeres da Costa C, Prodjinotho UF, Carabin H, Jackson E, Fleury A, Gabriel S, Ngowi BJ, Winkler AS. Efficacy and safety of antiparasitic therapy for neurocysticercosis in rural Tanzania: a prospective cohort study. Infection. 2023 Aug;51(4):1127-1139. doi: 10.1007/s15010-023-02021-y. Epub 2023 Mar 24. PMID 36961623
- See also: Efficacy and safety of antiparasitic therapy for neurocysticercosis in rural Tanzania: a prospective cohort study — http://link.springer.com/article/10.1007/s15010-023-02021-y